CLINICAL TRIAL: NCT06789003
Title: Evaluation of a PREHABilitation Protocol Using Adapted Physical Activity (APA) for Multiple Myeloma Patients Eligible for Intensive Autologous Stem Cell Transplantation Treatment (PREHAB-APA)
Brief Title: Evaluation of a PREHABilitation Protocol Using Adapted Physical Activity (APA) for Multiple Myeloma Patients Eligible for Intensive Autologous Stem Cell Transplantation Treatment
Acronym: PREHAB-APA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PREHAB-APA
Record Dates: First submitted 2025-01-06; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Adapted Physical Activity; Autologous stem cell transplantation; Quality of Life; Fatigue
MeSH Terms: conditions — Multiple Myeloma; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APA group (Experimental)
  Interventions: Other: Adapted exercises; Behavioral: Quality of Life questionnaire; Behavioral: Questionnaire of Fatigue; Behavioral: Physical activity questionnaire; Behavioral: Physical condition
- Control group (Active Comparator)
  Interventions: Other: No intervention; Behavioral: Quality of Life questionnaire; Behavioral: Questionnaire of Fatigue; Behavioral: Physical activity questionnaire; Behavioral: Physical condition

INTERVENTIONS:
Other: Adapted exercises — Patients will have 3 sessions a week: 1 strengthening session and 2 endurance sessions.
  For each session, patients will choose the exercises to be performed from the exercise booklet or the videos and records their observations in the patient notebook.
  Depending on the treatment plan, patients will have alternating supervised (in hospital) and unsupervised (at home) APA sessions, in order to follow the rhythm of their visits to the department.
  Each session will last 45 minutes with a medium intensity according to the Borg scale.
  Arms: APA group
Other: No intervention — Patients will not be practising adapted exercises as part of the study. They will be treated with chemotherapy according to standard practice.
  Arms: Control group
Behavioral: Quality of Life questionnaire — QoL questionnaire (EORTC QLQ-C30) at baseline, mid-term (after 2 cycles of chemotherapy), before transplantation, and after transplantation
Behavioral: Questionnaire of Fatigue — Questionnaire (EORTC QLQ-FA12) at baseline, mid-term (after 2 cycles of chemotherapy), before transplantation, and after transplantation
Behavioral: Physical activity questionnaire — Questionnaire (IPAQ) at baseline and after transplantation
Behavioral: Physical condition — Evaluation of physical condition at baseline, mid term (after 2 cycles of chemotherapy), before transplantation and after transplantation
  Other Names: 30s chair-stand test; Handgrip strength test; 6 minutes walk test

SUMMARY:
Adapted physical activity for patients with haematological malignancies generally has positive effects on quality of life, fatigue and physical condition. However, some studies show little or no effect.

This may be explained by inefficient protocols, but also by low rates of patient acceptability regarding the proposed exercises.

The multiplicity of APA protocols and the fluctuation of their results mean that validity, methodology and effects on patients need to be verified before they can be considered for implementation in healthcare services. A program must prove its feasibility, but patients must also adhere to it.

Acceptability can be measured by adherence, which represents the number of validated sessions in relation to the number of planned sessions, and by attrition, which corresponds to the number of stops or drop-outs for any reason. The various APA programs offered in the context of intensive auto or allograft treatment are limited, notably by adherence, which can fall by as much as 24%, and attrition, which can be as high as 67%. Optimization of the proposed exercises and follow-up methods is therefore necessary in order to propose an APA program that will be feasible, effective and acceptable to a maximum number of patients.

To meet these objectives for patients with multiple myeloma eligible for autologous stem cell transplantation, the protocol for this study took into consideration the various recommendations of previous publications and the guidelines from HAS (French National Authority for Health).

The ultimate goal of this study is to validate, in terms of effectiveness and acceptability, the methodology and in particular the use of new specific tools for optimizing an APA program. It will subsequently be offered to all patients with multiple myeloma eligible for autologous stem cell transplantation, independently of their age or physical condition, while respecting their rhythm and physical condition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* CML patient in chronic phase, eligible for oral therapy.
* Diagnosis of multiple myeloma.
* Patient eligible for autologous stem cell transplantation.
* Patient capable to read, understand and complete a questionnaire in french.
* WHO less than or equal to 2.
* Patient affiliated with french social security.
* Patient with a medical prescription for APA.

Exclusion Criteria:

* Patient with previous cancer within the previous 3 years (except basal cell and squamous cell skin cancers, carcinomas in situ of any type that have been previously resected, and stable prostate or breast cancers more than 3 years old and undergoing adjuvant hormone therapy).
* Medical contraindications to APA (heart failure, angina, unbalanced hypertension, bone metastases, severe osteoporosis, etc.)
* Sensory or motor neuropathy.
* Patient deprived of liberty, under guardianship or curatorship.
* Patient considered socially or psychologically unfit to be enrolled in a study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
1. Evaluate the effect of the APA program on fatigue status. | Baseline, mid-term assessment (after 2 cycles of chemotherapy, each cycle has a duration of 21 days), assessment before transplant and assessment after transplant (on average about 30 weeks after inclusion)
  Cancer Related Fatigue : EORTC QLQ-FA12 questionnaire (minimum = 0, maximum = 100, higher score means better outcome).

SECONDARY OUTCOMES:
Evaluate the effect of the APA program on quality of life. | Baseline, mid-term assessment (after 2 cycles of chemotherapy, each cycle has a duration of 21 days), assessment before transplant and assessment after transplant (on average about 30 weeks after inclusion)
  Quality of Life of Cancer Patients : EORTC QLQ-C30 questionnaire (minimum = 0, maximum = 100, higher score means better outcome).
Fitness assessment. | Baseline, mid-term assessment (after 2 cycles of chemotherapy, each cycle has a duration of 21 days), assessment before transplant and assessment after transplant (on average about 30 weeks after inclusion)
  6-minute walk test.
Fitness assessment. | Baseline, mid-term assessment (after 2 cycles of chemotherapy, each cycle has a duration of 21 days), assessment before transplant and assessment after transplant (on average about 30 weeks after inclusion)
  30-second chair-stand test.
Fitness assessment. | Baseline, mid-term assessment (after 2 cycles of chemotherapy, each cycle has a duration of 21 days), assessment before transplant and assessment after transplant (on average about 30 weeks after inclusion)
  Hand grip strength test.
Nutritional status. | Baseline, mid-term assessment (after 2 cycles of chemotherapy, each cycle has a duration of 21 days), assessment before transplant and assessment after transplant (on average about 30 weeks after inclusion)
  BMI.
Grade III-IV adverse events rate. | From inclusion to assessment after transplant (on average about 30 weeks after inclusion)
  According to Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Comparison of hospitalization length. | Assessment after transplant (on average about 30 weeks after inclusion)
  Hospitalization time (in days) after autologous stem cell transplantation.
15. Attraction to sport assessment. | Assessment after transplant (on average about 30 weeks after inclusion)
  IPAQ questionnaire (continuous score expressed as MET-min per week: MET level x minutes of activity/day x days per week, higher score means better outcome)
Adherence rate. | Assessment after transplant (on average about 30 weeks after inclusion)
  Percentage of patients who participated and validated more than 66 percent of the APA sessions recommended by the program.
Attrition rate. | Assessment after transplant (on average about 30 weeks after inclusion)
  Percentage of patients who discontinued the program during the course of the study among patients who received an autologous stem cell transplantation.
Rate of effective APA sessions. | Assessment after transplant (on average about 30 weeks after inclusion)
  Number of validated APA sessions divided by the number of planned sessions.
Reasons for discontinuing the APA program. | Assessment after transplant (on average about 30 weeks after inclusion)
  Self-reported reasons for discontinuation
Patient's comments and remarks. | 100 days after transplant
  Patient's follow-up notebook.
Patient satisfaction. | 100 days after transplant
  Satisfaction questionnaire. Likert-type scale (minimum = 0, maximum = 4, higher score means better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier d'Avignon, Hôpital Henri Duffaut, Avignon, France